CLINICAL TRIAL: NCT04330911
Title: The Effect of Supervised Exercise Programs on Exercise Capacity and Pulmonary Capacity in Type-2 Diabetic Patients
Brief Title: The Effects of Aerobic Exercises on Exercise Capacity in Type-2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emresenocak (Other)
Responsible Party: Sponsor-Investigator, Emresenocak, Research Assistant, Marmara University
Organization: Marmara University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2019.172
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Type-2 Diabetes
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: High-Intensity Interval Training Group (HIIT): The HIIT exercise protocol involved 28 minutes of treadmill efforts. The patients performed the interval training for 4 minutes with 80%HRmax and active recovery period maintained for 3 minutes with 60% HRmax on the treadmill with Karvonen formula.This protocol repeated 4 times in a session for 6 weeks.
  Moderate Intensity Continous Training (MICT): The MICT exercise protocol performed with %60 HRmax for 28 minutes for 6 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The HIIT Group (High Intensity Interval Training Group) (Experimental)
  Interventions: Procedure: Aerobic Exercise
- The MICT Group (Moderate Intensity Continous Training Group) (Experimental)
  Interventions: Procedure: Aerobic Exercise

INTERVENTIONS:
Procedure: Aerobic Exercise — Exercise loading is determined by increasing the heart rate. This loading calculated by Karvonen formulas (maximum %80 of Heart Rate)

SUMMARY:
Diabetes, beyond glycemic control, is a complex chronic disease that requires continuous medical care with multifactorial risk reduction strategies. It is necessary to reduce the likelihood of complications and additional problems that may develop in the long term. For this reason, guiding the patient to manage the disease process, equipping and supporting the patient with the necessary information is critical to prevent acute problems.

Exercise is the primary treatment method for diabetes patients. Exercise; It is the main treatment method used to increase aerobic capacity and improve respiratory capacity due to the positive effect it has on the body's structure and systems.

DETAILED DESCRIPTION:
Firstly, patients were examined by the specialist doctor. If patients appropriate for this study according to inclusion and exclusion criteria, they were consulted to Cardiologist for stress ECG test and acceptation report to high or moderate-intensity aerobic training.

After baseline testing (including aerobic capacity and lung capacity), appropriate patients were randomized to HIIT or MICT groups involving sixteenth sessions of exercise performed over 6 weeks The HIIT exercise protocol involved 28 minutes of treadmill efforts. The patients performed the interval training for 4 minutes with 80%HRmax and active recovery period maintained for 3 minutes with 60% HRmax on the treadmill. This protocol repeated 4 times in a session. The MICT exercise protocol performed with %60 HRmax for 28 minutes similarly HIIT group. A 10-min warm-up and 10-min cool-down period were included for all groups. All groups reassessed after the 6. weeks (end of the exercise program) and 12. weeks (follow-up period).

Aerobic capacity assessed with an Incremental Shuttle Walk Test (ISWT). Clinicians need to 10 m field, audiotape recorder, chronometer, and two markers. This test consists of 12 levels, every level maintains1 minute and the walking speed is increased after every1 minute intervals. If the patients wanted to stop because of fell breathless or can't reach the end of the 10 m line' last 0.5 m in the time allowed, the test was stopped.Estimated VO2max was calculated a formula as "Estimated VO2max (ml/dk/kg)= 4.19 + (0.025 x ISWT distance)".

The patient's pulmonary functions assessed with a digital spirometer (Pony FX, COSMED Inc., Italy). Spirometer device measures FVC, FEV1, FEV1/FVC and PEF values. During the test, upper extremity was straight and patients sitting straight position on the chair with their vertical feet on the floor. The measurements were performed 3 times and the best score recorded with mean and standard deviation.

The measurements were coded into the analysis program and checked by a second researcher.

Post-hoc power analysis was done using aerobic capacity data, which is the main output of our study. The power of the study was determined as 94%.

Patients who had missing data, patients who did not complete the 6-weeks exercise program and 12. weeks follow-up period were excluded from the analysis. All analyses were performed using the Statistical Package for the Social Sciences (SPSS) version 22. 0 for Windows. Data are expressed as mean ± standard deviation. The one-sample Kolmogorov-Smirnov test was performed to assess the distribution of data. Due to their distribution, numerical variables in different subjects were compared with the t-test or Mann-Whitney U test. Comparison of variables before and after the exercise program were compared by the paired t-test (parametric variable) or Wilcoxon test (non-parametric variable). Probability values were two-tailed, and a p-value of less than 0.05 was considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* patients with type-2 diabetes mellitus,
* patients who have sedentary lifestyle (<3 bouts of exercise per week and <30 minutes aerobic exercise period),
* non-smoking patients,
* not to lose more than 5% of total body weight in the last 6 months,
* blood pressure<160/100 mmHg

Exclusion Criteria:

* alcohol addiction in the last 12 months,
* patients who use insulin hormone,
* patients who have neuropathy or retinopathy,
* patients who have an acute cardiac event in the last 6 weeks,
* patients who have a disease at least 2 weeks in the last 1 month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Incremental Shuttle Walk Test-ISWT | Baseline Assessment
  Aerobic Capacity
Incremental Shuttle Walk Test-ISWT | End of the exercise period assessment (end of the 6. weeks)
  Aerobic Capacity
Incremental Shuttle Walk Test-ISWT | End of the follow-up period assessment (end of the 12. weeks)
  Aerobic Capacity
Digital Spirometer | Baseline Assessment
  FVC parameters were evaluated automatically.
Digital Spirometer | End of the follow-up period assessment (end of the 6. weeks)
  FVC parameters were evaluated automatically.
Digital Spirometer | End of the follow-up period assessment (end of the 12. weeks)
  FVC parameters were evaluated automatically.
Digital Spirometer | Baseline Assessment
  FEV1 were evaluated automatically.
Digital Spirometer | End of the follow-up period assessment (end of the 6. weeks)
  FEV1 were evaluated automatically.
Digital Spirometer | End of the follow-up period assessment (end of the 12. weeks)
  FEV1 were evaluated automatically.
Digital Spirometer | Baseline Assessment
  FEV1/FVC were evaluated automatically.
Digital Spirometer | End of the follow-up period assessment (end of the 6. weeks)
  FEV1/FVC were evaluated automatically.
Digital Spirometer | End of the follow-up period assessment (end of the 12. weeks)
  FEV1/FVC were evaluated automatically.
Digital Spirometer | Baseline Assessment
  PEF parameters were evaluated automatically.
Digital Spirometer | End of the follow-up period assessment (end of the 6. weeks)
  PEF parameters were evaluated automatically.
Digital Spirometer | End of the follow-up period assessment (end of the 12. weeks)
  PEF parameters were evaluated automatically.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No